CLINICAL TRIAL: NCT04819243
Title: Randomized Phase II Study of Talazoparib Versus Talazoparib Plus Atezolizumab After Palbociclib Combination Endocrine Therapy for Patients with Premenopausal HR+/HER2- Metastatic Breast Cancer Harboring HRD Scar
Brief Title: PALbociclib Endocrine Therapy Followed by Talazo Vs. Talazoz-Atezo Study
Acronym: Young-PALETTA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Yeon Hee Park, Clinical Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-01-075
Record Dates: First submitted 2021-03-25; First posted 2021-03-26 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Premenopausal HR+/HER2- Metastatic Breast Cancer
MeSH Terms: interventions — talazoparib; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Atezolizumab+Talazoparib (Experimental): 1. st line treatment
     * Palbociclib 125mg po D1-21
     * AI : Prescribed as per local guideline
     * GnRH agonist: Prescribed as per local guideline (or ET + CDK4/6 inhibitors + GnRH agonist)
  2. nd line treatment
     * Talazoparib 1mg po
     * Atezolizumab 1200mg IV (3week)
  Interventions: Drug: Pabociclib, Endocrine(or ET + CDK4/6 inhibitors), Talazoparib, Atezolizumab
- Talazoparib (Experimental): 1. st line treatment
     * Palbociclib 125mg po D1-21
     * AI : Prescribed as per local guideline
     * GnRH agonist: Prescribed as per local guideline (or ET + CDK4/6 inhibitors + GnRH agonist)
  2. nd line treatment - Talazoparib 1mg po
  Interventions: Drug: Pabociclib, Endocrine(or ET + CDK4/6 inhibitors), Talazoparib,

INTERVENTIONS:
Drug: Pabociclib, Endocrine(or ET + CDK4/6 inhibitors), Talazoparib, Atezolizumab — * Palbociclib 125mg
  * AI
  * GnRH agonist (or ET + CDK4/6 inhibitors + GnRH agonist)
  * Talazoparib
  * Atezolizumab
  Arms: Atezolizumab+Talazoparib
Drug: Pabociclib, Endocrine(or ET + CDK4/6 inhibitors), Talazoparib, — * Palbociclib 125mg
  * AI
  * GnRH agonist (or ET + CDK4/6 inhibitors + GnRH agonist)
  * Talazoparib
  Arms: Talazoparib

SUMMARY:
This study is a prospective, two-arm, randomized phase II study of talazoparib versus talazoparib plus atezolizumab in ER+ premeonopausal women with metastatic breast cancer harboring HRD scar

1st line treatment: GnRH agonist + Aromatase Inhibitor(AI) + Palbociclib 28 days after the last treatment of 1st line treatment(., randomization for 2nd line treatment is conducte to arm A(Talazoparib+Atezolizumab) and arm B(Talazoparib monotherapy)

DETAILED DESCRIPTION:
1. st line treatment

   * Palbociclib: A capsule will be administered once a day for 21 days and rest for 7 days (1cycle=28days)
   * AI treatment: D1~28 days. Take once a day. Prescribed according to local prescribe guideline.
   * GnRH agonist: At D1 for every cycle with 4 week (+3days) interval via subcutaneous injection.

   (or ET + CDK4/6 inhibitors + GnRH agonist)
2. nd line treatment

28 days after the last treatment of 1st line treatment, randomization for 2nd line treatment is conducte to arm A(Talazoparib+Atezolizumab) and arm B(Talazoparib monotherapy)

* Talazoparib: Take orally once a day at the same time
* Atezolizumab: 1,200mg, at D1 of each cycle. Applicable for arm A only.

ELIGIBILITY:
* Eligibility criteria prior to 1L treatment:

  1. Histologically confirmed metastatic breast cancer with or without measurable disease
  2. Patients who have stage IV breast cancer at diagnosis (de novo) or have progressed on distant metastatic sites after curative surgery: locally advanced disease not amenable to distant metastasis are eligible as well as disease with distant metastasis
  3. Confirmed germline pathogenic BRCA1 and/or 2 mutation or 35 HRD-related gene alterations (see Appendix 16.5)
  4. age > 19 years
  5. ECOG performance status 0 - 2
  6. Patient has HER2 IHC0, IHC1+, or ICH2+/ISH-, as determined according to ASCO/CAP guidelines breast cancer
  7. Patient has ER positive and/or PgR positive according to American Society of Clinical Oncology/College of American Pathologists (ASCO/CAP) guidelines, defined as 1% of tumor cells stained positive based on the most recent tumor biopsy and assessed locally
  8. Female patients should be premenopausal. Premenopausal status is defined as either:

     A. Patient had last menstrual period within the last 12 months B. If on tamoxifen within the past 3 months, with a plasma estradiol ≥10 pg/mL and FSH ≤40 IU/l or in the premenopausal range, according to local laboratory definition C. in case of chemotherapy induced amenorrhea, with a plasma estradiol ≥10 pg/mL) and/or FSH ≤40IU/l or in the premenopausal range according to local laboratory definition.
  9. Patient with treatment history as bellows:

     A. In patients with de novo metastatic breast cancer(who had stage IV disease at first diagnosis of breast cancer), B. In patients with recurrent metastatic breast cancer, recurrence during or after completion or discontinuation of adjuvant endocrine therapy (regardless of the treatment free interval) are eligible.

     C. One line of prior cytotoxic chemotherapy(except platinum based chemotherapy) in metastatic breast cancer is permitted.
  10. No possibility of pregnancy and/or urine or serum beta-HCG negative
  11. Adequate bone marrow function (≥ ANC 1,500/ul, ≥ platelet 100,000/ul, ≥ Hemoglobin 9.0 g/dl)
  12. Adequate renal function (≤ serum creatinine 1.5 mg/dl or CCr ≥ 60 ml/min)
  13. Adequate liver function (≤ serum bilirubin 2.0 mg/dl, ≤ AST/ALT x 3 upper normal limit). If the subject has liver metastasis, AST/ALT x 5 upper normal limit is acceptable.
  14. Patients who were already established on bisphosphonate therapy or denosumab may continue.
  15. Patients agreed to use effective contraception or not of childbearing potential
  16. Written informed consent
  17. Patients agreed to offer tumor tissue and blood for biomarker analysis
* Exclusion criteria prior to 1L treatment

  1. Postmenopausal women except women who had BSO (Bilateral Salpingo Oophorectomy)
  2. Serious uncontrolled intercurrent infections within 4 weeks prior to Cycle 1 Day 1 of 1st Treatment
  3. Serious intercurrent medical or psychiatric illness, including active cardiac disease
  4. Participants who are pregnant or breast feeding or intending to become pregnant during the study or within 5 months after the final dose of study treatments.
  5. Second primary malignancy(except in situ carcinoma of the cervix or adequately treated nonmelanomatous carcinoma of the skin or favorable thyroid papillary carcinoma(follicular thyroid cancer, including PTC) or other malignancy treated at least 5 years previously with no evidence of recurrence)
  6. Patients has received previous endocrine treatments in the metastatic setting (Except tamoxifen only ± GnRH agonist)
  7. Patients has received previous aromatase inhibitor (less than 1 year after the last dose)
  8. Patients has received previous treatment with CDK 4/6 inhibitors, OR PARP1 inhibitors, OR immune check point inhibitors (less than 1 year after the last dose)
  9. Known brain metastases, symptomatic or asymptomatic
  10. History of clinically significant liver disease, current alcohol abuse or known active infection
  11. History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus (SLE), rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis
  12. Prior allogeneic stem cell or solid organ transplantation
  13. History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia (i.e. bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest computerised tomography (CT) scan
  14. Active tuberculosis
  15. Receipt of a live, attenuated vaccine within 4 weeks prior to Cycle 1 Day 1 of 1st Treatment or anticipation that a live, attenuated vaccine will be required during atezolizumab treatment or within 5 months after the last dose of atezolizumab
  16. Treatment with systemic immunostimulatory agents (including but not limited to interferons or interlukin [IL]-2) within 4 weeks or five half-lives of the drug (whichever is longer) prior to Cycle 1 Day 1 of 1st Treatment
  17. Treatment with systemic corticosteroids or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, mycophenolate, and anti-tumour necrosis factor [TNF] agents) within 2 weeks prior to Cycle 1 Day 1 of 1st Treatment, or anticipated requirement for systemic immunosuppressive medications during the trial
* Inclusion criteria prior to 2L treatment

  * For subjects who were enrolled in the 1L treatment part of the study, inclusion criteria 1)-4) should be met.
  * For subjects who were not enrolled in the 1L treatment part of the study, all of the following inclusion criteria should be met prior to the study enrollment.

    1. ECOG performance status 0 - 2
    2. Adequate bone marrow function (≥ANC 1,500/ul, ≥platelet 100,000/ul, ≥Hemoglobin 9.0 g/dl)
    3. Adequate renal function (≤ serum creatinine 1.5 mg/dl or CCr ≥ 60 ml/min)
    4. Adequate liver function (≤ serum bilirubin 2.0 mg/dl, ≤ AST/ALT x 3 upper normal limit) If the subject has liver metastasis, AST/ALT x 5 upper normal limit is acceptable
    5. Histologically confirmed metastatic or locally advanced breast cancer that is not amenable to curative surgery, with or without measurable disease. Patients who have stage IV breast cancer at diagnosis (de novo) or have progressed on distant metastatic sites after curative surgery are eligible.
    6. Prior treatment with endocrine-based therapy + CDK4/6 inhibitor for metastatic or inoperable locally advanced breast cancer. Allowed endocrine-based therapy is as below:

       A. Aromatase Inhibitor B. For subjects who had disease progression during or after the adjuvant aromatase inhibitor therapy, fulvestrant C. Up to one line of chemotherapy for metastatic or inoperable locally advanced breast cancer is allowed except for platinum based chemotherapy.
    7. Confirmed germline pathogenic BRCA1 and/or BRCA2 mutation or 35 HRD-related gene alterations (see Appendix 16.5)
    8. age > 19 years
    9. Patient has HER2 IHC0, IHC1+, or ICH2+/ISH-, as determined according to ASCO/CAP guidelines breast cancer
    10. Patient has ER positive and/or PgR positive according to American Society of Clinical Oncology/College of American Pathologists (ASCO/CAP) guidelines, defined as 1% of tumor cells stained positive based on the most recent tumor biopsy and assessed locally
    11. Female patients should be premenopausal. Premenopausal status is defined as either:

        A. Patient had last menstrual period within the last 12 months B. If on tamoxifen within the past 3 months, with a plasma estradiol ≥10 pg/mL and FSH ≤40 IU/l or in the premenopausal range, according to local laboratory definition C. in case of chemotherapy induced amenorrhea, with a plasma estradiol ≥10 pg/mL) and/or FSH ≤40IU/l or in the premenopausal range according to local laboratory definition.

        D. If the subject started ovarian function suppression, above A-C criteria should be met prior to starting ovarian function suppression.
    12. No possibility of pregnancy and/or urine or serum beta-HCG negative
    13. Patients may continue an ongoing bisphosphonate or denosumab therapy.
    14. Patients who agreed to use an effective contraception method or have no childbearing potential
    15. Written informed consent
    16. Patients who agreed to offer tumor tissue and blood for biomarker analysis
* Exclusion criteria prior to 2L treatment

  * For subjects who participate only in the 2L treatment part of the study, all exclusion criteria should be met prior to study enrollment.

    1. Postmenopausal women except women who had BSO (Bilateral Salpingo Oophorectomy)
    2. Serious intercurrent medical or psychiatric illness, including active cardiac disease
    3. Participants who are pregnant or breast feeding or intending to become pregnant during the study or within 5 months after the final dose of study treatments.
    4. Second primary malignancy(except in situ carcinoma of the cervix or adequately treated nonmelanomatous carcinoma of the skin or favorable thyroid papillary carcinoma(follicular thyroid cancer, including PTC) or other malignancy treated at least 5 years previously with no evidence of recurrence)
    5. Patients who have previously received PARP1 inhibitors OR immune check point inhibitors
    6. Patients who have previously received platinum based chemotherapy or two or more lines of chemotherapy for metastatic or inoperable locally advanced breast cancer
    7. Known brain metastases, symptomatic or asymptomatic
    8. History of clinically significant liver disease, current alcohol abuse or known active infection
    9. History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus (SLE), rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis
    10. Prior allogeneic stem cell or solid organ transplantation
    11. History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia (i.e. bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest computerised tomography (CT) scan
    12. Active tuberculosis
    13. Receipt of a live, attenuated vaccine within 4 weeks prior to Cycle 1 Day 1 of 1st Treatment or anticipation that a live, attenuated vaccine will be required during atezolizumab treatment or within 5 months after the last dose of atezolizumab
    14. Treatment with systemic immunostimulatory agents (including but not limited to interferons or interlukin [IL]-2) within 4 weeks or five half-lives of the drug (whichever is longer) prior to Cycle 1 Day 1 of 1st Treatment
    15. Treatment with systemic corticosteroids or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, mycophenolate, and anti-tumour necrosis factor [TNF] agents) within 2 weeks prior to Cycle 1 Day 1 of 1st Treatment, or anticipated requirement for systemic immunosuppressive medications during the trial

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2021-08-25 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
2nd Progression free survival (PFS) | The time until the time of the first event(the progression of a recorded disease of breast cancer or death from all causes) in 2nd line treatment. Up to 72months
  To assess measures of clinical efficacy. It is a measure of the period of survival without disease progression by Kaplan-Meier method.

SECONDARY OUTCOMES:
Composite PFS (1st PFS + 2nd PFS) | The time from the day 1 of first therapy to the time of first event (documented disease progression of breast cancer or death due to any cause) in 1st and 2nd line therapy. Up to 72months
  To assess measures of clinical efficacy. It is a measure of the period of survival without disease progression by Kaplan-Meier method.
Overall survival (OS) | Survival will be measured as the time from the randomization occurs after Progression of 1st line to the date of death. Up to 72months
  To assess secondary measures of clinical efficacy.
Toxicity assessment | from the date of informed consent signature to 28 days after last drug administration
  Clinical and laboratory toxicity/symptomatology will be graded based on the NCIC CTG v5.0
Quality of Life (QoL) | from the date of informed consent signature to 28 days after last drug administration
  The QoL will be evaluated using EQ5D

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung medical Center, Seoul, Gannam-gu, South Korea

IPD SHARING:
Plan to Share IPD: No